CLINICAL TRIAL: NCT05277142
Title: EFFECT OF NEUROMUSCULAR ELECTRICAL STIMULATION ON DYSPHAGIA IN CHILDREN WITH DOWN SYNDROME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Walid Saber Hussain, assistant lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7689
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): they received oral motor training for 40 minutes 3 times/week for twelve successive weeks.
  Interventions: Other: oral motor training
- Group (B) (Experimental): They received the same Oral motor training program of Group A for 20 minutes in addition to Neuromuscular Electrical Stimulation (NMES) at intensity ranged from (3-5mA) duration for 20 minutes and frequency of 80 HZ 3 times/week for twelve successive weeks.
  Interventions: Other: oral motor training; Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: oral motor training — they received oral motor training for 40 minutes 3 times/week for twelve successive weeks.
Device: Neuromuscular Electrical Stimulation — They received the same Oral motor training program of Group A for 20 minutes in addition to Neuromuscular Electrical Stimulation (NMES) at intensity ranged from (3-5mA) duration for 20 minutes and frequency of 80 HZ 3 times/week for twelve successive weeks
  Arms: Group (B)

SUMMARY:
Although some western studies have been conducted to determine the nature of eating problems and oral motor training in children with Down syndrome, these studies are limited. Most of the studies were done in Down syndrome infants. Since feeding is a skill that develops by 2 years of age and refines till 6 years of age (Delaney & Arvedson 2008), it is essential to study the children in this age group as well. Moreover, there is a dearth of studies investigating the impact of oral motor exercises on feeding problems of the child, which may, in turn, hinder the progress of the child during the intervention. Blissett J., (2018) reported that the behaviours of both caretaker, therapist and infant during feeding contribute significantly to the overall success of the feeding interaction as well as feeding performance. Parents/caregivers play an important role in feeding the child, as they have the first-hand exposure and experience in feeding their child, awareness of the child's feeding behaviours, likes and dislikes of food and communication behaviour during hunger. Consequently, they are the best people to describe their child's feeding problems. Hence, this study involves the administration of a scale on the parent/caregiver to elicit information about the physical, functional and emotional aspects of drooling. Such studies in the Egyptian context are limited. The paucity of literature makes it clear that there are deeper underlying complex issues about oral motor exercises in children with Down syndrome that needs to be investigated. The in-depth assessment and treatment of oral motor skills will provide valuable input to the physical therapists during the treatment of feeding problems in children with Down syndrome. This would help the therapist and clinician in planning and prioritizing the goals during therapy. The information will also help in counselling the caregivers, deciding the success or failure of feeding therapy and thereby help in predicting the prognosis of the child.

ELIGIBILITY:
Inclusion Criteria:

* 1- Their age ranged from 3 to 6 years. 2- Both genders were included. 3- The participating children having the ability to understand and follow simple instructions (IQ level not less than 50).

  4- They did not have any visual or auditory problems. 5- They did not be treated with special medications affecting mental functions. 6- They had score from 4 to 7 according to functional oral intake scale.

Exclusion Criteria:

* 1- Children with history of epilepsy. 2- Children with dental deformities. 3- Children with chest infections or unstable cardiac status. 4- Children with infective skin conditions. 5- Children with gum disorders.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
1- Oral Motor Assessment Scale | 12 weeks
  The Oral Motor Assessment Scale (OMAS) are used as an outcome measurement in intervention studies. The scale items were elaborated by a multidisciplinary team comprising dentists and speech therapists. It TEMPhas characteristics dat differentiate it from other scales coz it does not require dat the subject obey commands and it does not include speech assessment
2- Pediatric Eating Assessment Tool- Pedi EAT | 12 weeks
  Teh Pediatric Eating Assessment Tool (PediEAT) measures symptoms of feeding problems in young children. Content validity was established using DeVellis' methods of scale development (13) through systematic item generation and evaluation by clinical and research experts as well as by teh intended respondents: parents of children both with and without feeding problems
3- Pediatric Eating Assessment Tool | 12 weeks
  The Pediatric Version of the Eating Assessment Tool (PEDI-EAT-10) is the pediatric version of the 10-item Eating Assessment Tool (EAT-10), which is a reliable and valid dysphagia symptom specific outcome tool The Eating Assessment Tool-10 (EAT-10) is a validated, commonly used tool in clinical practice, which serves for the assessment of symptom-specific outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Emad, Giza, Egypt